CLINICAL TRIAL: NCT03117478
Title: The Impact of Meditation Practice on Attention and Emotion Regulation :Studies on Neural Correlation in Brain Imagery and Biomarkers of Stress and Inflammation
Brief Title: Brain and Mindfulness
Acronym: MEDITATION
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 69HCL16_0678
Record Dates: First submitted 2017-02-08; First posted 2017-04-18 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Healthy
MeSH Terms: interventions — Meditation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- 1. Participants without meditation experience (Other): Novices. Note that there is no meditation intervention in this study but that the two groups differ in their lifetime meditation experience.
  Interventions: Other: Magneto-encephalography (MEG); Other: Electro-encephalography (EEG); Other: Functional Magnetic Resonance Imaging (fMRI); Other: Anatomical Magnetic Resonance Imaging (aMRI); Other: Meditation
- 2. Participant with a significant meditation experience (Other): Experts : > 5000 hours of practice during their life. Note that there is no meditation intervention in this study but that the two groups differ in their lifetime meditation experience.
  Interventions: Other: Magneto-encephalography (MEG); Other: Electro-encephalography (EEG); Other: Functional Magnetic Resonance Imaging (fMRI); Other: Anatomical Magnetic Resonance Imaging (aMRI); Other: Meditation
- 3. Participants without meditation experience (Other): Novices. There is no meditation intervention during the study but the investigators investigate the effects of meditation by comparing 2 groups who differ in their life time meditation experience (i.e., novices vs. experts).
  Interventions: Other: Magneto-encephalography (MEG); Other: Electro-encephalography (EEG); Other: Functional Magnetic Resonance Imaging (fMRI); Other: Anatomical Magnetic Resonance Imaging (aMRI)
- 4. Participant with a significant meditation experience (Other): Experts : > 5000 hours of practice during their life. There is no meditation intervention during the study but the investigators investigate the effects of meditation by comparing 2 groups who differ in their life time meditation experience (i.e., novices vs. experts).
  Interventions: Other: Magneto-encephalography (MEG); Other: Electro-encephalography (EEG); Other: Functional Magnetic Resonance Imaging (fMRI); Other: Anatomical Magnetic Resonance Imaging (aMRI)

INTERVENTIONS:
Other: Magneto-encephalography (MEG) — Magneto-encephalography
Other: Electro-encephalography (EEG) — Electro-encephalography
Other: Functional Magnetic Resonance Imaging (fMRI) — Functional Magnetic Resonance Imaging
Other: Anatomical Magnetic Resonance Imaging (aMRI) — Anatomical Magnetic Resonance Imaging
Other: Meditation — Meditation
  Arms: 1. Participants without meditation experience; 2. Participant with a significant meditation experience

SUMMARY:
The main aim of this project is to explore the neuro-anatomical and -physiological correlates of meditation on attention and emotion-regulation. By investigating this, our scientific goal is to more generally identify the mechanisms and biomarkers of health and mental well-being. Therefore, the investigators use non-invasive imaging like Magneto-EncephaloGraphy (MEG), ElectroEncephaloGraphy (EEG), functional and anatomic Magnetic Resonance Imaging (MRI; including Diffusion tensor - DTI). These brain measures will then be linked to behavioral measurements. Experimental methods (i.e., simple computer tasks) will be used to measure attention, conscious perception and regulation of pain and emotion.

ELIGIBILITY:
Inclusion Criteria:

* Age : 25-70
* Being affiliated to a social security system.
* Motivated to participate in this study.

Exclusion Criteria:

* Medication acting on the central nervous system
* Opioids, Antidepressive Agents.
* Actual or previous neurological or psychiatric illnesses
* Chronic pain or any other medical condition which is related to pain or an increased sensitivity to pain.
* Not having a personal or family history of epilepsy
* Alcohol or drugs consumption 2 days before or during the study.

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 169 (Actual)
Dates: Start 2016-03-19 (Actual); Primary Completion 2019-10-16 (Actual); Study Completion 2019-10-16 (Actual)

PRIMARY OUTCOMES:
Anatomical MRI scan | Day 1
  Brain structure
Functional MRI scan | Day1
  Brain activation: Haemodynamic response - BOLD signal.
EEG | Day 1
  Event-related potential fields : amplitude in fT and latency in ms. Oscillations : power spectral density and time-frequency oscillations in fT^2/Hz

SECONDARY OUTCOMES:
Behavioral measure : Accuracy of the performed task actions | Day 1
  Participants will perform behavioral computer tasks in which accuracy and speed is important. Performance behavior will be measured in this task: Accuracy of the performed task actions: number of errors and hits
Psychophysics: Pain threshold | Day 1
  Pain threshold: The threshold of pain or pain threshold is the point along a curve of increasing perception of a stimulus at which pain begins to be felt. The temperature in degrees Celcius at which heat becomes painful for a recipient.
Psychophysiology : Respiration | Day 1
  Respiration rate: breaths/minute
Subjective experience of the participant | Day 1
Studies biomarkers of inflammation | Day 1
  area of the inflamed site in mm^2, obtained by automatic image processing of a photography
Behavioral measure : Speed of the performed task actions | Day 1
  Participants will perform behavioral computer tasks in which accuracy and speed is important. Performance behavior will be measured in this task: Speed of the performed task actions: in ms.
Psychophysiology : Heart | Day 1
  Heart Rate: pulses/minute
Psychophysiology : Heart rate variability | Day 1
  Heart rate variability (HRV): Using an electrocardiogram, the variation in the beat-to-beat interval; measured in ms.
Psychophysiology : Muscles | Day 1
  Electromyography (EMG): Recording the electrical activity produced by muscles; measured in mV.
Psychophysiology : Eyes | Day 1
  Eye gaze position: relative to center of the screen, in imm
Psychophysiology : Pupillar response | Day 1
  Pupillar response: pupil diameter, in mm.
Electrogastrogram | Day 1
  Recording the electrical signals that travel through the stomach muscles and control the muscles' contractions (waves/minute)

CONTACTS AND LOCATIONS:
Overall Officials: Sandrine SONIE, MD, Principal Investigator — Le Vinatier
Locations (1):
- Le Vinatier, Bron, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zorn J, Abdoun O, Sonie S, Lutz A. Cognitive Defusion Is a Core Cognitive Mechanism for the Sensory-Affective Uncoupling of Pain During Mindfulness Meditation. Psychosom Med. 2021 Jul-Aug 01;83(6):566-578. doi: 10.1097/PSY.0000000000000938. PMID 33790200
- [Background] Zorn J, Abdoun O, Bouet R, Lutz A. Mindfulness meditation is related to sensory-affective uncoupling of pain in trained novice and expert practitioners. Eur J Pain. 2020 Aug;24(7):1301-1313. doi: 10.1002/ejp.1576. Epub 2020 May 7. PMID 32311185
- [Background] Poublan-Couzardot A, Lecaignard F, Fucci E, Davidson RJ, Mattout J, Lutz A, Abdoun O. Time-resolved dynamic computational modeling of human EEG recordings reveals gradients of generative mechanisms for the MMN response. PLoS Comput Biol. 2023 Dec 13;19(12):e1010557. doi: 10.1371/journal.pcbi.1010557. eCollection 2023 Dec. PMID 38091350
- [Background] Poletti S, Abdoun O, Zorn J, Lutz A. Pain regulation during mindfulness meditation: Phenomenological fingerprints in novices and experts practitioners. Eur J Pain. 2021 Aug;25(7):1583-1602. doi: 10.1002/ejp.1774. Epub 2021 Apr 22. PMID 33797842
- [Background] Katyal S, Abdoun O, Mounier H, Lutz A. Reduced processing of afforded actions while observing mental content as ongoing mental phenomena. Sci Rep. 2024 May 2;14(1):10130. doi: 10.1038/s41598-024-60934-6. PMID 38698150
- [Background] Fucci E, Poublan-Couzardot A, Abdoun O, Lutz A. No effect of focused attention and open monitoring meditation on EEG auditory mismatch negativity in expert and novice practitioners. Int J Psychophysiol. 2022 Jun;176:62-72. doi: 10.1016/j.ijpsycho.2022.03.010. Epub 2022 Mar 28. PMID 35358612
- [Background] Fucci E, Abdoun O, Lutz A. Auditory perceptual learning is not affected by anticipatory anxiety in the healthy population except for highly anxious individuals: EEG evidence. Clin Neurophysiol. 2019 Jul;130(7):1135-1143. doi: 10.1016/j.clinph.2019.04.010. Epub 2019 Apr 27. PMID 31085447
- [Background] Fucci E, Abdoun O, Baquedano C, Lutz A. Ready to help, no matter what you did: Responsibility attribution does not influence compassion in expert Buddhist practitioners. J Exp Psychol Gen. 2024 Apr;153(4):1093-1111. doi: 10.1037/xge0001542. Epub 2024 Feb 22. PMID 38386366
- [Background] Czajko S, Zorn J, Daumail L, Chetelat G, Margulies DS, Lutz A. Exploring the Embodied Mind: Functional Connectome Fingerprinting of Meditation Expertise. Biol Psychiatry Glob Open Sci. 2024 Aug 9;4(6):100372. doi: 10.1016/j.bpsgos.2024.100372. eCollection 2024 Nov. PMID 39309211
- [Background] Abdoun O, Zorn J, Poletti S, Fucci E, Lutz A. Training novice practitioners to reliably report their meditation experience using shared phenomenological dimensions. Conscious Cogn. 2019 Feb;68:57-72. doi: 10.1016/j.concog.2019.01.004. Epub 2019 Jan 15. PMID 30658238